CLINICAL TRIAL: NCT01605032
Title: Phase II Study Assessing the Efficacy and Toxicity of PK--directed Intravenous Busulfan in Combination With High--Dose Melphalan and Bortezomib as Conditioning Regimen for First--Line Autologous Hematopoietic Stem Cell Transplantation in Patients With Multiple Myeloma
Brief Title: Busulfan, Melphalan, and Bortezomib Before First-Line Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ira Braunschweig, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-12-434; NCI-2013-01207 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-102; 11-12-434 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2012-03-07; First posted 2012-05-24 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Busulfan; Melphalan; Bortezomib; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (busulfan, melphalan, bortezomib, autologous PBSCT) (Experimental): CONDITIONING: Patients receive busulfan IV over 3 hours on days -6 to -3, melphalan IV over 20 minutes on day -2, and bortezomib IV over 3-5 seconds on days -6, -3, 1, and 4.
  TRANSPLANT: Patients undergo autologous PBSCT on day 0.
  Interventions: Drug: Busulfan; Drug: Melphalan; Drug: Bortezomib; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: Busulfan — Given IV
Drug: Melphalan — Given IV
  Other Names: Alkeran
Drug: Bortezomib — Given IV
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: Autologous Stem Cell Transplantation
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation

SUMMARY:
This phase II trial studies how well busulfan, melphalan, and bortezomib before first-line stem cell transplant works in treating patients with multiple myeloma. Giving chemotherapy before a peripheral blood stem cell transplant may stop the growth of cancer cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood and stored. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response rate as defined by the International Myeloma Working Group (IMWG) criteria for patients with multiple myeloma treated with high dose chemotherapy with pharmacokinetic (PK) directed intravenous (IV) busulfan, bortezomib and melphalan (Bu/BTZ/Mel140) followed by autologous hematopoietic stem cell transplantation (ASCT) as first line therapy.

SECONDARY OBJECTIVES:

I. To determine the overall response rate of the regimen Bu/BTZ/Mel140. II. To determine the treatment related toxicity and mortality of the regimen, including 100-day mortality rates.

III. To determine the duration of response, time to progression, progression-free survival, event-free survival and overall survival for this conditioning regimen.

IV. To determine whether there is a gender or race difference in the pharmacokinetic profile of IV busulfan.

V. To determine methylation and gene expression signatures of pre-treatment bone marrow plasma cells and explore associations of these signatures with outcome.

OUTLINE:

CONDITIONING: Patients receive busulfan IV over 3 hours on days -6 to -3, melphalan IV over 20 minutes on day -2, and bortezomib IV over 3-5 seconds on days -6, -3, 1, and 4.

TRANSPLANT: Patients undergo autologous peripheral blood stem cell transplant (PBSCT) on day 0.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed multiple myeloma
* Measurable disease must be present as defined by protein criteria (quantifiable M-component in serum, urine or serum free light chains) in order to evaluate response as per IMWG; non-secretory patients are eligible provided the patient has > 20% plasmacytosis OR multiple (> 3) focal plasmacytomas or focal lesions on magnetic resonance imaging (MRI)
* Patients must have received induction chemotherapy for myeloma, but not more than 12 months of prior chemotherapy for this disease, and must be eligible for the first planned autologous transplant
* A minimum stem cell dose of 2.0 x 10^6 cluster of differentiation 34-positive (CD34+) cells/kg has been collected
* Life expectancy of greater than 12 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL (unless myeloma related)
* Absolute neutrophil count >= 1,500/mcL (unless myeloma related)
* Platelets >= 50,000/mcL (unless myeloma related)
* Total bilirubin =< 2 x institutional upper limit of normal unless 2nd to Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Ejection fraction by echocardiogram (ECHO) or multi gated acquisition scan (MUGA) >= 40% performed within 60 days prior to registration
* Patients must have adequate pulmonary function studies: > 50% of predicted on mechanical aspects (forced expiratory volume in one second [FEV1], forced vital capacity [FVC]) and diffusion capacity (diffusing capacity of the lung for carbon monoxide [DLCO]) > 50% of predicted, within 60 days of registration; if the patients is unable to complete pulmonary function tests due to multiple myeloma (MM) related pain or condition, exception may be granted if the principal investigator (PI) documents that the patient is a candidate for high dose therapy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least six months following the stem cell transplantation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Prior treatment history of autologous hematopoietic stem cell transplant (HSCT) or high-dose chemotherapy with stem cell rescue for any medical reason, not limited to myeloma treatment
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to or other agents used in the study, such as busulfan, melphalan, bortezomib, boron, or mannitol
* Grade 2 or greater peripheral neuropathy within 14 days prior to enrollment
* Unresolved grade >= 3 non-hematologic toxicity from previous therapy; patients with grade 2 toxicity will be eligible at the discretion of the PI
* Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ; cancer treated with curative intent < 5 years will not be allowed unless approved by the PI; cancer treated with curative intent > 5 years will be allowed
* Patients must not have significant co-morbid medical condition
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients must not have suffered recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with busulfan
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients found to have an active hepatitis B infection (hepatitis B surface antigen +) are not eligible unless they meet ONE of the following criteria:

  * Patient is able to start dual anti-hepatitis (Hep) B therapy prior to enrollment with adefovir and telbivudine
  * Patient is already on dual anti-hepatitis B therapy
  * Consultation and co-management with a hepatitis expert regarding hepatitis B treatment is strongly encouraged before and during the trial
* Patients, who are positive for hepatitis B core antibody, but negative for the hepatitis B surface antigen, should be started on lamivudine 100 mg daily until at least 3 months post stem cell transplant

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Braunschweig, Principal Investigator — Albert Einstein College of Medicine
Locations (4):
- United States (4):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Cancer Institute, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT): CONDITIONING: Patients receive busulfan IV over 3 hours on days -6 to -3, melphalan IV over 20 minutes on day -2, and bortezomib IV over 3-5 seconds on days -6, -3, 1, and 4.
  TRANSPLANT: Patients undergo autologous PBSCT on day 0.
  Busulfan: Given IV
  Melphalan: Given IV
  Bortezomib: Given IV
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous PBSCT
  Peripheral Blood Stem Cell Transplantation: Undergo autologous PBSCT
Period: Overall Study
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
Started | 19
Completed | 18
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
Number analyzed (Participants) | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [32 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ISS stage at diagnosis [Number; unit: participants] — The international staging system (ISS) was used to stage the patients.
  * Stage I: Serum beta-2 microglobulin < 3.5 mg/L and serum albumin ≥3.5 g/dL - Good outcome
  * Stage II: Not stage I or stage III - Slightly worse outcome
  * Stage III: Serum beta-2 microglobulin ≥ 5.5 mg/L - Worse outcome
  For 16 of them ISS was available at initial diagnosis.
  participants
    Stage 1 | 4
    Stage 2 | 7
    Stage 3 | 5
    Stage unkown | 3
Cytogenetics/FISH at diagnosis [Number; unit: participants]
  High risk | 2
  Intermediate risk | 2
  Standard risk | 6
  Unknown | 10
Previous treatment [Number; unit: participants]
  Bortezomib-containing regimen | 17
  Immunomodulatory agent-containing regimen | 7
Response before ASCT [Count of Participants; unit: Participants]
  Complete response | 1
  Very Good partial response | 2
  Partial response | 10
  Stable disease | 5
  Progressive disease | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response as Determined by the IMWG Criteria
Description: Number of patients achieved complete response after the treatment regimen
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
Number analyzed (Participants) | 19
Participants | 2

2. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
Number analyzed (Participants) | 19
Participants
  Complete response | 2
  Partial response | 17

3. Secondary Outcome: Mortality
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
Number analyzed (Participants) | 19
Participants | 1

4. Secondary Outcome: Time-to-progression
Time Frame: From start of treatment to disease progression with deaths, up to 2 years
Population: The outcome measure 'Time to Progression' was not collected
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Description: The progression free survival was assessed over a period of 2 years
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
Number analyzed (Participants) | 19
Participants | 11

6. Secondary Outcome: Overall Survival
Description: The overall survival of patients was measured of a period of 2 years.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
Number analyzed (Participants) | 19
Participants | 18

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT)
All-Cause Mortality (participants affected / at risk) | 1/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT) (N=19)
Death - 70 days after the autologous stem cell transplant (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Busulfan, Melphalan, Bortezomib, Autologous PBSCT) (N=19)
Electrolyte abnormalities (General disorders) | 17 — Grade 3 & 4
Oral mucositis (Gastrointestinal disorders) | 18 — Grade 3 & 4
Dysphagia/Odynophagia (Gastrointestinal disorders) | 17 — Grade 3 & 4
Transaminitis (Endocrine disorders) | 13 — Grade 3 & 4
Nausea and/or vomitting (Gastrointestinal disorders) | 18 — Grade 3 & 4
Diarrhea (Gastrointestinal disorders) | 15 — Grade 3 & 4
Abdominal pain (Gastrointestinal disorders) | 3 — Grade 3 & 4
Fever without neutropenia (General disorders) | 4 — Grade 3 & 4
Febrile neutropenia (Immune system disorders) | 14 — Grade 3 & 4
Infections (Infections and infestations) | 8 — Grade 3, 4 & 5
Noninfectious pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 2 — Grade 3 & 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT01605032/Prot_SAP_000.pdf
  • Informed Consent Form (2014-04-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT01605032/ICF_001.pdf